CLINICAL TRIAL: NCT05406570
Title: Personalized Tidal Volume According to Cardiopulmonary Interactions in ARDS
Brief Title: Personalized Tidal Volume in ARDS (VT4HEMOD)
Acronym: VT4HEMOD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 69HCL21_1272; 2021-A02996-35 (Other: ANSM)
Record Dates: First submitted 2022-06-02; First posted 2022-06-06 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-11

CONDITIONS: Acute Respiratory Distress Syndrome
Keywords: Acute Respiratory Distress Syndrome; cardiopulmonary interaction; tidal volume; computed tomography
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standardized tidal volume (Active Comparator): Ventilation with tidal volume 6 ml/kg
  Interventions: Procedure: Standardized ventilation; Procedure: Personalized ventilation
- Personalized tidal volume (Experimental): Ventilation with tidal volume aiming to minimize cardiopulmonary interactions as assessed by pulse pressure variation
  Interventions: Procedure: Standardized ventilation; Procedure: Personalized ventilation

INTERVENTIONS:
Procedure: Standardized ventilation — Patient will be ventilated with tidal volume 6 mL/kg predicted body weight (PBW) and positive end-expiratory pressure (PEEP) according to the PEEP-FiO2 table of the ARMA trial. A CT scan will be performed with this ventilatory setting and the patients will be switched to the other group
Procedure: Personalized ventilation — Patient will be ventilated with PEEP according to the PEEP-FiO2 table of the ARMA trial. Tidal volume will be selected as the tidal volume minimizing cardiopulmonary interactions as assessed on arterial pressure tracing, during a VT trial. A CT scan will be performed with this ventilatory setting and the patients will be switched to the other group.

SUMMARY:
Treatment of acute respiratory distress syndrome (ARDS) relies on invasive mechanical ventilation with supposedly protective settings (low tidal volume ventilation). Mortality of ARDS remains high in observational studies (40 to 50%). Approximately 30% of ARDS patients exhibit tidal hyperinflation despite low tidal volume ventilation, suggesting that personalization of tidal volume is required to improve ARDS prognostic. To date, reliable bedside tools to adjust tidal volume are lacking. Excessive tidal volume can be detected using computed tomography by quantification of tidal hyperinflation, but this technique is reserved to research studies and requires patient transport to imaging facility.

Mechanical ventilation generates cardio-pulmonary interaction, whose magnitude is influenced by tidal volume and respiratory system characteristics. Pulse pressure variation is a bedside tool with potential to quantify cardio-pulmonary interactions. Increasing tidal volume will decrease right ventricular preload and increase right ventricular afterload, hence maximizing cardio-pulmonary interactions.

The investigators hypothesize that pulse pressure variation might help to detect excessive tidal volume during a tidal volume challenge (i.e. stepwise increase in tidal volume)

ELIGIBILITY:
Inclusion Criteria:

1. Age greater then 18 years old
2. ARDS according to the BERLIN definition with PaO2/FiO2 ratio ≤ 150 mm Hg
3. invasive mechanical ventilation in volume controlled mode with tidal volume set to 6 ml/kg predicted body weight
4. use of sedation and neuromuscular-blocking agents
5. arterial catheter allowing computation of pulse contour cardiac output calibrated with thermodilution
6. central venous catheter implanted in the superior vena cava territory
7. esophageal balloon
8. Computed tomography planned by attending physician

Exclusion Criteria:

1. Previous inclusion in current study
2. Acute cor pulmonale
3. ECMO
4. Arterial pH < 7.21 despite respiratory rate set to a maximum of 35/min
5. Pneumothorax or bronchopleural fistula
6. Decision to withdraw or withhold life sustaining treatment with 24 hours from inclusion
7. Contra-indication of transport to imaging facility
8. Intracranial hypertension
9. Tricuspid or pulmonary mechanical valve
10. Tricuspid or pulmonary infective endocarditis
11. Pace maker with intracardiac leads
12. Right ventricle tumor
13. Complete left bundle block
14. Intrathoracic metallic device
15. COPD
16. Cardiac arrythmia
17. Vesical pressure > 15 mm Hg
18. Lower limb amputation
19. Inferior vena cava thrombosis
20. Patient under an exclusion period relative to participation to another clinical trial
21. Patient under a legal protective measure
22. Patient not affiliated to social security
23. lac of patient/representative consent
24. Pregnancy
25. Breast feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2022-12-29 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Tidal hyperinflation | 5 minutes - This endpoint will be assessed 5 minutes after ventilatory adjustment
  Difference between hyperinflated volume in computed tomography images acquired at end-inspiration (defined by the volume of voxels with CT-number < -900) and hyperinflated volume in computed tomography images acquired at end-expiration (defined by the volume of voxels with CT-number < -900). This difference will be standardized to predicted body weight using the formula of the ARMA trial.

SECONDARY OUTCOMES:
Tidal volume | 5 hours - This endpoint will be assessed through study completion (approximately 4-5 hours after study inclusion)
  Standardized versus personalized tidal volume

CONTACTS AND LOCATIONS:
Locations (1):
- Hospices Civils de Lyon - Hôpital de la Croix Rousse - Service de Médecine Intensive Réanimation, Lyon, France

IPD SHARING:
Plan to Share IPD: Undecided